CLINICAL TRIAL: NCT00005223
Title: Epidemiology of APO- and Lipoproteins in Elderly Women
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1102; R29HL040489 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2001-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

SUMMARY:
To examine the complex interactions among the traditional cardiovascular risk factors, particularly lipoprotein and apoprotein levels, genetic and other characteristics, and lifestyle habits in elderly women.

DETAILED DESCRIPTION:
BACKGROUND:

Coronary heart disease is the leading cause of death in both men and women 65 years of age and older, and in 1982, it was estimated that it accounted for about 32.4 percent of all deaths in this age group and may have contributed to death in an additional 12.1 percent. Coronary heart disease mortality rates increase steeply with age, even in those over 65 years of age. Death rates for males continue to be higher than females although the sex ratio declined sharply with age. Data from Framingham suggest that although the incidence of coronary heart disease rises with age in both males and females, the incidence rate rises more steeply in elderly females compared with elderly males. Despite the magnitude of this problem, in 1988 the majority of the knowledge on coronary heart disease and its risk factors related to the disease in middle-aged persons--primarily males. More information was needed about coronary heart disease and its risk factors in elderly women. Also, the atherosclerotic process develops over many years and the risk factors which relate to the evolution of atherosclerosis are highly correlated within an individual. Therefore, it is likely that risk factors, such as lipoproteins and apoproteins will be important determinants of coronary heart disease in older persons primarily because of this observed correlation within individuals over time, and their long-term association with the development and progression of atherosclerosis. In addition, identification of the high risk individual is a goal of many epidemiologic investigations. It is possible that qualitative examination of the polymorphisms of the apoproteins could in fact assist in the identification of women at high risk of coronary heart disease who are in need of aggressive prophylaxis. These genetic markers represent a second generation of risk factors for coronary heart disease.

DESIGN NARRATIVE:

The study was ancillary to the multicenter Study of Osteoporotic Fractures (SOF), a prospective study on risk factors for hip and wrist fractures supported by the National Institute of Arthritis and Musculoskeletal and Skin Diseases. The cross-sectional study involved a sample of subjects at the Pittsburgh Center. The distribution and interrelationships of lipoproteins and apoproteins were described as were their relationships to age, years since menopause, type of menopause, and lifestyle factors such as physical activity, alcohol consumption, cigarette smoking, obesity, and use of estrogens/progestins. The frequency of phenotypes of the polymorphisms of apoprotein A-IV and E were examined to determine whether these phenotypes were associated with specific patterns of lipo- and apoproteins. The hypothesis was tested that the degree to which lifestyle characteristics explain the variability in lipoproteins and apoproteins depended on the genetic makeup of the individual.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-04; Study Completion 1993-03 (Actual)

REFERENCES:
- [Background] Vogt MT, Cauley JA, Kuller LH, Nevitt MC. Bone mineral density and blood flow to the lower extremities: the study of osteoporotic fractures. J Bone Miner Res. 1997 Feb;12(2):283-9. doi: 10.1359/jbmr.1997.12.2.283. PMID 9041062
- [Background] Vogt MT, Cauley JA, Kuller LH. Apolipoprotein E phenotype, arterial disease, and mortality among older women: the study of osteoporotic fractures. Genet Epidemiol. 1997;14(2):147-56. doi: 10.1002/(SICI)1098-2272(1997)14:23.0.CO;2-4. PMID 9129960
- [Background] Vogt MT, Nevitt MC, Cauley JA. Back problems and atherosclerosis. The Study of Osteoporotic Fractures. Spine (Phila Pa 1976). 1997 Dec 1;22(23):2741-7. doi: 10.1097/00007632-199712010-00008. PMID 9431608
- [Background] Cauley JA, Gutai JP, Kuller LH, Powell JG. The relation of endogenous sex steroid hormone concentrations to serum lipid and lipoprotein levels in postmenopausal women. Am J Epidemiol. 1990 Nov;132(5):884-94. doi: 10.1093/oxfordjournals.aje.a115731. PMID 2239903
- [Background] Vogt MT, Cauley JA, Kuller LH, Nevitt MC. Functional status and mobility among elderly women with lower extremity arterial disease: the Study of Osteoporotic Fractures. J Am Geriatr Soc. 1994 Sep;42(9):923-9. doi: 10.1111/j.1532-5415.1994.tb06581.x. PMID 8064098
- [Background] Danielson ME, Cauley JA, Rohay JM. Physical activity and its association with plasma lipids and lipoproteins in elderly women. Ann Epidemiol. 1993 Jul;3(4):351-7. doi: 10.1016/1047-2797(93)90061-8. PMID 8275210
- [Background] Cauley JA, Gutai JP, Glynn NW, Paternostro-Bayles M, Cottington E, Kuller LH. Serum estrone concentrations and coronary artery disease in postmenopausal women. Arterioscler Thromb. 1994 Jan;14(1):14-8. doi: 10.1161/01.atv.14.1.14. PMID 8274469
- [Background] Carson CA, Cauley JA, Caggiula AW. Relation of caffeine intake to blood lipids in elderly women. Am J Epidemiol. 1993 Jul 15;138(2):94-100. doi: 10.1093/oxfordjournals.aje.a116839. PMID 8342534
- [Background] Vogt MT, Cauley JA, Newman AB, Kuller LH, Hulley SB. Decreased ankle/arm blood pressure index and mortality in elderly women. JAMA. 1993 Jul 28;270(4):465-9. PMID 8320785
- [Background] Cauley JA, Eichner JE, Kamboh MI, Ferrell RE, Kuller LH. Apo E allele frequencies in younger (age 42-50) vs older (age 65-90) women. Genet Epidemiol. 1993;10(1):27-34. doi: 10.1002/gepi.1370100104. PMID 8472931
- [Background] Vogt MT, Cauley JA, Kuller LH, Hulley SB. Prevalence and correlates of lower extremity arterial disease in elderly women. Am J Epidemiol. 1993 Mar 1;137(5):559-68. doi: 10.1093/oxfordjournals.aje.a116709. PMID 8465807
- [Background] Ganguli M, Cauley JA, DeKosky ST, Kamboh MI. Dementia among elderly apolipoprotein E type 4/4 homozygotes: a prospective study. Genet Epidemiol. 1995;12(3):309-11. doi: 10.1002/gepi.1370120308. PMID 7557352
- [Background] Cauley JA, Zmuda JM, Yaffe K, Kuller LH, Ferrell RE, Wisniewski SR, Cummings SR. Apolipoprotein E polymorphism: A new genetic marker of hip fracture risk--The Study of Osteoporotic Fractures. J Bone Miner Res. 1999 Jul;14(7):1175-81. doi: 10.1359/jbmr.1999.14.7.1175. PMID 10404018